CLINICAL TRIAL: NCT03648710
Title: Community Health Workers and Mobile Health for Emerging Adults Transitioning Sickle Cell Disease Care
Brief Title: Community Health Workers and mHealth for Sickle Cell Disease Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: St. Christopher's Hospital for Children (Other); Children's Hospital Medical Center, Cincinnati (Other); Steven and Alexandra Cohen Children's Medical Center (Individual); Connecticut Children's Medical Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-015106
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (No Intervention): Enhanced usual care will be standardized across sites with transition/transfer of care checklists that will be used at all sites. Enhanced usual care will minimally include (1) patient seen by the pediatric provider with the parent outside the examination room, (2) a social work consult to screen and address sociodemographic risk factors, (3) information on health insurance adequacy provided to patient, (4) adult hematologist identified, (5) adult primary care provider identified, (6) medical release signed, and (7) medical record viewable or sent to adult provider.
- Peer Community Health Worker (Experimental): The CHW program will primarily be modeled after the highly successful IMPaCT Program developed by the Penn Center for Community Health Workers and CHOP's Youth CHW Program for Pediatric to Adult Transitions developed by our research team, which were both developed with high levels of patient input. SCD specific content and expertise from the CHW Program through the Sickle Cell Disease Association of American Philadelphia Delaware Valley Chapter and other published models will be included. Components will include: 1) development of patient-centered goals and individualized action plan around self-care, symptom tracking, and transition to adult care; 2) provision of information, skills, and tips; and 3) tailored peer support using telephone calls and/or visits
  Interventions: Other: Peer Community Health Worker
- Mobile Health (Experimental): All participants enrolled in the mHealth arm will download an enhanced version of iManage, which was developed by Co-Investigator Lori Crosby at and adolescents and young adult patients with SCD. Components include: 1) development of patient-centered goals around self-care, symptom tracking, and transition to adult care; 2) provision of information, skills, and tips; 3) virtual peer support where users can encourage others to complete goals, forms teams, and interact with other youth with SCD; and 4) daily symptom tracking and visual tracking of goal completion. Investigators will add with daily tailored texting.
  Interventions: Other: Mobile Health

INTERVENTIONS:
Other: Peer Community Health Worker — Participants will be communicating with their CHWs on a weekly basis, which is consistent with other successful community health worker protocols with published efficacy. Community Health Workers will be peers with sickle cell disease, who have successfully transitioned and are under 30 years of age.
  Arms: Peer Community Health Worker
Other: Mobile Health — A mobile health application created as a resource for young adults transitioning.
  Arms: Mobile Health

SUMMARY:
This study will compare the effectiveness of two self-management support interventions-Community Health Workers (CHW) and mobile health (mHealth)-versus enhanced usual care to improve health-related quality of life and acute care use for transitioning youth with sickle cell disease (SCD), and identify and quantify mediators and moderators of intervention treatment effects.

DETAILED DESCRIPTION:
Emerging adults with sickle cell disease (SCD) experience a seven-fold increase in mortality rates during the transition period (16-25 years of age). This staggering increase in mortality and acute care utilization during this vulnerable period is partly due to difficulty coordinating care during the transition to adult care. Critical psychosocial issues further compound the vulnerability of emerging adults with SCD during the transition from pediatric to adult care9. Unfortunately, none of these transition intervention studies included adolescents or young adults with SCD. Patients, parents, and providers of those with SCD agree that the ability to independently perform chronic disease self-management is critical to staying healthy during this turbulent transition period.

Self-management support is a key component of the Chronic Care Model. Community health worker (CHW) programs are increasingly popular and have efficacy on chronic disease self-management and system navigation. Mobile health platforms are equally popular, and have efficacy on self-management and adherence. Unfortunately, the effectiveness of mHealth and tailored texting among emerging adults with SCD is still unknown. Furthermore, also unknown is the comparative effectiveness of CHW programs and mHealth.

The purpose of the study is to determine the comparative effectiveness of CHW programs and mHealth among emerging adults with SCD during transition versus enhanced usual care to improve health-related quality of life and acute care use for transitioning youth with SCD.

The primary objective of this study is to compare the effectiveness of two self-management support interventions (community health workers and mobile health) versus enhanced usual care to improve health-related quality of life and acute care use for transitioning youth with SCD. The secondary objectives are to:

* Identify and quantify whether patient activation, self-management behaviors, biologic markers, and transfer to adult care are mediators of intervention treatment effects.
* Identify individual and family factors that moderate intervention treatment effects

The exploratory aim is to:

•Explore the association of enhancements to usual care on pediatric and adult acute utilization

The study population will consist of all patients with SCD who are 17 or older and are appropriate for transfer to an adult hematologist within 12 months. Excluded are individuals with an intellectual disability that is severe enough that the individual would not have the capacity to interact with a mobile or web-based program even with assistance or have a conversation with a community health worker (i.e. non-verbal).

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 17 years or older
* Have sickle cell disease, defined as those individuals with HbSS, HbSC, HbSβ0Thal, HbSβ+Thal genotypes
* Receive care at a participating pediatric sickle cell disease center.
* Appropriate for transfer to an adult hematologist within 12 months

Exclusion Criteria:

* Individuals with an intellectual disability that is severe enough that the individual would not have the capacity to interact with a mobile or web-based program even with assistance or have a conversation with a community health worker (i.e. non-verbal). Individuals without access to a mobile device, tablet or computer.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (HRQOL) | Baseline, 6 months, 12months, and 18 months.
  Health-Related Quality of life will be assessed with the PedsQL Sickle Cell Disease (SCD) Module. The PedsQL Sickle Cell Disease Module is a well-validated for use in adolescents and young adults with chronic disease and use a Likert response scale, with higher scores indicating better HRQOL and lower SCD symptoms and problems. The PedsQL SCD Module is a 43-item that measures nine scales: Pain and Hurt (9 items), Pain Impact (10 items), Pain Management and Control (2 items), Worry I (5 items), Worry II (2 items), Emotions (2 items), Treatment (7 items), Communication I (3 items), and Communication II (3 items).

SECONDARY OUTCOMES:
Sickle cell disease knowledge | Baseline, 6months, 12 months, 18 months
  Measured using the Sickle Cell Disease Knowledge Questionnaire (SCDKQ). SCDKQ is a 20-item survey. All questions have answer choices of true or false.
Transition Readiness | Baseline, 6 months, 12 months, 18 months
  Measured using the Transition Readiness Assessment Questionnaire (TRAQ). TRAQ is a 20 item survey of transition readiness. Answer choices are based on stages of change and are on a 5-point scale.
Social Support | Baseline, 6 months, 12 months, 18 months
  Measured using the Medical Outcomes Study Social Support Survey (MOS-SSS). The MOS-SSS is a 19-item survey. Answer choices are on a 5-point Likert scale ranging from "none of the time" to "all of the time".
Coping skills | Baseline, 6 months, 12 months, 18 months
  Coping strategies using the Coping Strategies Questionnaire (Brief COPE). The Brief COPE is a 28-item survey with answer choices on a 4-point Likert scale, ranging from "I haven't been doing this at all" to "I've been doing this a lot".
Education and vocational planning | Baseline, 6 months, 12 months, 18 months
  Using the Transition Intervention Program - Readiness for Transition (TIPS-RFT) sub scale to measure education and vocational planning. The educational and vocational planning subscale of the TIPS-RFT is a 4 question subscale.
Quality of care received | Baseline, 6 months, 12 months, 18 months
  Using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) measure. The quality of care received subscale is from the ASCQ-Me. The subscale is 27 multiple choice questions.
Medical Adherence Scale | Baseline, 6 months, 12 months, 18 months
  Medication adherence will be measured using the Medical Adherence Measure (MAM). The MAM is a 17 question multiple choice survey.

CONTACTS AND LOCATIONS:
Overall Officials: David Rubin, MD, Principal Investigator — Children's Hospital of Philadelphia; Sophia Jan, MD, Principal Investigator — Cohen's Children Medical Center/Northwell Health; Kim Smith-Whitley, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Cohen's Children's Medical Center, New Hyde Park, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christophers Hospital for Children, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Jan S, Steinway C, Belton T, Shults J, Bennett L, Teng O, Griffis H, Aygun B, Appiah-Kubi A, Apollonsky N, Boruchov D, Niss O, Schwartz L, Crosby L, Barakat L, Andemariam B, Mulchan SS, Rubin D, Smith-Whitley K. Community Health Worker and Mobile Health Interventions for Quality of Life Among Young Adults With Sickle Cell Disease: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2543571. doi: 10.1001/jamanetworkopen.2025.43571. PMID 41247734
- [Derived] Belton TD, Steinway CM, Teng O, Shults J, Barakat LP, Aygun B, Appiah-Kubi A, Crosby LE, Niss O, Andemariam B, Schwartz LA, Luma S, Smith KA, Johnson TB, Rubin DM, Smith-Whitley KM, Jan S. The Community Health Workers and Mobile Health for Emerging Adults Transitioning Sickle Cell Disease Care (COMETS) Trial: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 4;14:e69239. doi: 10.2196/69239. PMID 40905609
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077